CLINICAL TRIAL: NCT06200350
Title: Personalized Recommendation System of Specific Challenges for Sport Activities: Practical Approach to Football
Brief Title: Personalized Recommendation System for Sport Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Juan López Barreiro, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09-181223; ED481A-2021/350 (Other Grant/Funding Number: Xunta de Galicia)
Record Dates: First submitted 2023-12-27; First posted 2024-01-11 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Health Behavior
Keywords: Performance; Football; Recommender system; Training; Gamification; Blockchain; NFT; Reward
MeSH Terms: conditions — Health Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Control group will continue with the conventional training. Experimental group will carry out a tailored training based on the profile of each participant.
Who Masked: Outcomes Assessor
Masking Description: As this study needs a intervention different from the conventional, the blinding of the participants is imposible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group will carry out the tailored training proposed by de recommender system, and followed and encouraged by the blockchain dApp.
  Interventions: Other: Experimental group
- Control group (Active Comparator): This group will continue with the traditional training planned.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Tailored training based on the profile of each participant.
  Arms: Experimental group
Other: Control group — They will continue with the traditional training.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to test and compare the effects of a tailored algorithm recommendation of sport activities concreted in challenges to improve some critical performance dimensions.

Q1: Improving participant performance is achieved by using personalized sports activity recommendation using an algorithm and tracking compliance using a decentralized application (dApp)? Q2: Are participants satisfied with the performance and simplicity of the dApp used?

Participants will be asked to do specific activities recommended by the developed recommender system. The activities to be carried out will be conditioned by the profile obtained from each participant at the beginning of the intervention. They will consist of reinforcement activities for the dimensions with the lowest scores.

Researchers will compare a experimental group and a control group to see if the dimensions assessed at the beginning of the intervention were improved.

ELIGIBILITY:
Inclusion Criteria:

* Amateur football players.
* Aged between 14 and 18 years old.
* Without any injury.
* The ones who can attend the assessing sessions and fill in the informed consent form.

Exclusion Criteria:

* Aged different from the indicated above.
* Injured.
* Missing one of the assessing sessions.
* Not performing the proposed training twice, or not registering two or more training sessions.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Score of the system usability at the end of the intervention | At the end of the intervention (8 weeks)
  System Usability Scale is a scale from 0 to 100 points to assess the usability of the system used in the intervention.

SECONDARY OUTCOMES:
Squat Jump (SJ) | At baseline and after 8 weeks
  Lower body capacity assessed using the SJ
Abdominal planck (AP) | At baseline and after 8 weeks
  Core capacity assessed using the abdominal plank lasting time
Push ups (PU) | At baseline and after 8 weeks
  Upper body capacity assessed using the number of pushups performed in one minute
Cooper Test (GE) | At baseline and after 8 weeks
  General endurance assessed using the Cooper Test
15m sprint (SE-15) | At baseline and after 8 weeks
  Special endurance assessed using the 15m sprint
Countermovement Jump (CMJ) | At baseline and after 8 weeks
  Special endurance assessed using the CMJ

OTHER OUTCOMES:
Sociodemographic outcomes | At baseline
  Body weight, height, age and gender.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vigo, Pontevedra, Pontevedra, Spain